CLINICAL TRIAL: NCT04775238
Title: Metallic Nanoparticles: Evaluation of Their Antibacterial, Antibiofilm and Synergistic Effect in Combination With Antibiotics on Nosocomial Bacteria
Brief Title: Effect of Metallic Nanoparticles on Nosocomial Bacteria
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Nahed Fathallah Fahmy, lecturer of medical microbiology & immunology departement -faculty of medicine- sohag university, Sohag University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Soh-Med-21-02-21
Record Dates: First submitted 2021-02-22; First posted 2021-03-01 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-02

CONDITIONS: Nosocomial Infections
Keywords: Staphylococcus aureus; Pseudomonas; silver nanoparticles; copper nanoparticles
MeSH Terms: conditions — Cross Infection; Staphylococcal Infections; Pseudomonas Infections | interventions — colloidal silver

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Staphylococcus aureus) (Active Comparator): Staphylococcus aureus is an example of gram positive bacteria which is a strong biofilm producer and highly resistant to antibiotics. Staphylococcus aureus will be exposed to silver nanoparticles and copper nanoparticles separately to study their antibacterial and biofilm inhibiting properties and their synergistic effect in combination with antibiotics.
  Interventions: Other: Silver nanoparticles; Other: Copper nanoparticles
- Group 2 (Pseudomonas aeruginosa ) (Active Comparator): Pseudomonas aeruginosa is an example of gram negative bacteria which is a strong biofilm producer and highly resistant to antibiotics. Pseudomonas aeruginosa will be exposed to silver nanoparticles and copper nanoparticles separately to study their antibacterial and biofilm inhibiting properties and their synergistic effect in combination with antibiotics.
  Interventions: Other: Silver nanoparticles; Other: Copper nanoparticles

INTERVENTIONS:
Other: Silver nanoparticles — AgNPs (19±5 nm)
  Other Names: AgNPs
Other: Copper nanoparticles — CuNPs (150-350 nm)
  Other Names: CuNPs

SUMMARY:
This research aims to study the properties of metallic nanoparticles"MNPs" (silver nanoparticles "AgNps" and copper nanoparticles "CuNps") on the 2 most common nosocomial bacteria which are highly resistant to antibiotics including Staphylococcus aureus and Pseudomonas aeruginosa, to evaluate the growth inhibiting properties of MNPs on all bacterial isolates, to evaluate the biofilm inhibitory effect on biofilm forming bacterial isolates and the synergistic effect of these MNPs in combination with antibiotics on the antibiotic resistant isolates.

DETAILED DESCRIPTION:
There is a rapid increase in the number of health care associated infections (HAIs) due to multi-drug resistant (MDR) bacterial strains which have a worse prognosis being associated with significant morbidity and mortality, particularly in critically ill patients. The main problem with MDR strains is their limited treatment options, posing a major challenge for health care providers.The increasing utilization and immense studies of nanoparticles have brought new perspectives towards new antimicrobial material that could hinder the MDR bacteria pandemic currently faced. Particularly, metallic nanoparticles exhibit strong biocidal properties on different bacterial species, including MDR bacteria. Another important aspect of the antimicrobial properties of metallic nanoparticles is their potential to eradicate or inhibit microbial biofilm formation, which is an important virulence factor in many localized chronic infections.

ELIGIBILITY:
Inclusion Criteria:

* Urinary tract infections (UTI)
* Surgical site infections (SSI)
* Catheter related blood stream infection (CRBSI)
* Infected burns
* Chest infection

Exclusion Criteria:

* Patients less than 18 years.
* Community acquired infections

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-02-27 (Actual); Primary Completion 2021-06-20 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Measurement of the inhibition zone diameter by (mm) around wells containing silver nanoparticles on nutrient agar containing 105 cfu/ml (colony forming unit/ml) Staphylococcus aureus | 24 hours
  Well diffusion method
Measurement of the inhibition zone diameter by (mm) around wells containing silver nanoparticles on nutrient agar containing 105 cfu/ml Pseudomonas | 24 hours
  Well diffusion method
Measurement of the inhibition zone diameter by (mm) around wells containing copper nanoparticles on nutrient agar containing 105 cfu/ml Staphylococcus aureus | 24 hours
  disc diffusion method
Measurement of the inhibition zone diameter by (mm) around wells containing copper nanoparticles on nutrient agar containing 105 cfu/ml Pseudomonas | 24 hours
  disc diffusion method
Antibiofilm Activity:12 μg/mL of AgNPs will be added to 107 CFU/mL of Staph aureus. using a microtiter plate reader at 595 nm, biofilm scores: nonbiofilm forming (-), weak (+), moderate (++), and strong (+++) | 24 hours
  Modified Tissue Culture Plate method (TCP):by ELISA
Antibiofilm Activity:12 μg/mL of CuNPs will be added to 107 CFU/mL of Staph aureus. using a microtiter plate reader at 595 nm, biofilm scores: nonbiofilm forming (-), weak (+), moderate (++), and strong (+++) | 24 hours
  Modified Tissue Culture Plate method (TCP):by ELISA
Antibiofilm Activity:12 μg/mL of AgNPs will be added to 107 CFU/mL of Pseudomonas. Using a microtiter plate reader at 595 nm, biofilm scores: nonbiofilm forming (-), weak (+), moderate (++), and strong (+++) | 24 hours
  Modified Tissue Culture Plate method (TCP):by ELISA
Antibiofilm Activity:12 μg/mL of CuNPs will be added to 107 CFU/mL of Pseudomonas. Using a microtiter plate reader at 595 nm, biofilm scores: nonbiofilm forming (-), weak (+), moderate (++), and strong (+++) | 24 hours
  Modified Tissue Culture Plate method (TCP):by ELISA
Synergism with antibiotics: cefoxitin, Tetracyclin, Ciprofloxacin, Rifampin, Linezolide impregnated with 42.5 μg/mL AgNPs will be placed on nutrient agar containing 105 cfu/ml of Staph aureus. Inhibition zones will be measured (mm). | 24 hours
  disc diffusion method
Synergism with antibiotics: cefoxitin, Tetracyclin, Ciprofloxacin, Rifampin, Linezolide impregnated with 85 μg/mL CuNPs will be placed on nutrient agar containing 105 cfu/ml of Staph aureus. Inhibition zones will be measured (mm). | 24 hours
  disc diffusion method
Synergism with antibiotics:piperacillin-tazobactam, Aztreonam, Imipenem, Colistin, Ciprofloxacin impregnated with 42.5 μg/mL AgNPs will be placed on nutrient agar containing 105 cfu/ml of Pseudomonas. Inhibition zones will be measured (mm). | 24 hours
  disc diffusion method
Synergism with antibiotics:piperacillin-tazobactam, Aztreonam, Imipenem, Colistin ,Gentamicin, Ciprofloxacin impregnated with 85 μg/mL CuNPs will be placed on nutrient agar containing 105 cfu/ml of Pseudomonas. Inhibition zones will be measured (mm). | 24 hours
  disc diffusion method

CONTACTS AND LOCATIONS:
Overall Officials: Nahed Fathallah, lecturer, Principal Investigator — Sohag University
Locations (1):
- Faculty of medicine - sohag university, Sohag, Egypt